CLINICAL TRIAL: NCT02883751
Title: Effects of Phototherapy on the Healing of Ulcers Following Minor Lower Extermity Amputations in Patients With Diabetes Mellitus - Protocol for a Randomized, Controlled, Double-blind, Clinical Trial
Brief Title: Phototherapy in DM Amputation Ulcers.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI is no longer working at UniNove
Sponsor: University of Nove de Julho (Other)
Collaborators: Daniela de Fátima Teixeira da Silva (Unknown); Monica Ribeiro Ventura (Unknown)
Responsible Party: Principal Investigator, Cristiane Miranda Franca, Professor at the Biophotonics applied to Health Sciences Post Graduation Program, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1.464.664
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Mellitus; Amputation Stumps; Diabetic Foot
Keywords: diabetes mellitus; amputation stumps; diabetic foot; phototherapy; clinical trial
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot | interventions — Low-Level Light Therapy; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Active Comparator): Control group - gold standard: Conventional ulcer treatment with Rayon® and essential fatty acids (Dersani®). Cleaning of the surgical wound will be performed with saline solution. The wound will then be covered with a sterile polyethylene film, over which the LED plate will be positioned for placebo treatment (emission of sound, but with the device switched off). After 10 minutes, the LED plate and polyethylene film will be removed and the surgical wound will be covered with rayon moistened with essential fatty acids (following the standard protocol of the hospital), followed by the application of gauze and finalization with a crepe bandage.
  Interventions: Procedure: Control group
- LED group (Experimental): LED group: Cleaning of the surgical wound will be performed with saline solution and the wound will be covered with a sterile polyethylene film, over which the LED plate will be positioned for active treatment with the device switched on. After 10 minutes, the LED plate and polyethylene film will be removed and the surgical wound will be covered with rayon moistened with essential fatty acids (following the standard protocol of the hospital), followed by the application of gauze and finalization with a crepe bandage.
  Interventions: Radiation: LED

INTERVENTIONS:
Radiation: LED — A device with 36, rectangular, red LEDs, registered with the Brazilian National Health Surveillance Agency (ANVISA authorization nº 8.04554.6), λ = (650 ± 20) nm, with an output power of 324 mW and an output area of 2.54 cm2 (Cosmedical, Brazil), will be enveloped with sterile, disposable, plastic wrap (transparent in the red wavelength) to permit contact with the skin for ten minutes during each session. The plastic wrap will be changed after each use. The amount of energy delivered will be 194.4 J.
  Other Names: Photobiomodulation with light emmiting diode (LED)
  Arms: LED group
Procedure: Control group — Conventional ulcer treatment with rayon® (Polar Fix, Polar Fix, Mauá, SP, Brazil) and essential fatty acids (Dersani®, Saniplan, Daudt, São Paulo, SP, Brazil) (composition: decanoic acid, caprylic acid, hexanoic acid, lauric acid, linoleic acid, lecithin, retinyl palmitate, tocopheryl acetate and alpha-tocopheryl).
  Arms: Control group

SUMMARY:
Diabetes mellitus is a major public health problem and it is estimated that 300 million individuals will be affected by the year 2030. Non-diabetic ulcers are one of the most frequent complications of this disease and, if untreated, can lead to the amputation of lower limbs. Thus, there has been growing interest in the use of light emitting diode (LED) devices to accelerate the tissue repair process and lower the cost of ulcer treatment in this population. The Mandaqui hospital complex is a general, tertiary, teaching hospital that is a reference center for revascularization surgery and endovascular treatment in Brazil. The aim of the proposed study is to evaluate the action of LED therapy on the complete healing of ulcers following minor amputations in patients with Diabetes mellitus. Methods: A single-center, randomized, controlled, double-blind, clinical trial with two parallel groups will be conducted following the criteria of the CONSORT Statement. The project will be registered with www.clinicaltrials.gov. The sample will be composed of 40 patients with a diagnosis of Diabetes mellitus in follow up at the vascular clinic of Mandaqui hospital complex who meet the inclusion criteria. The control group (n = 20) will receive traditional rayon bandages with essential fatty acids and secondary coverage with gauze, which will be changed on a weekly basis. The treatment group (n = 20) will be submitted to LED therapy (635 nm; 4 J/cm2; 10 minutes) with weekly applications and the ulcers will also receive the traditional bandage treatment described above. The patients will be followed up until the complete closure of the ulcer, which will be the primary outcome. The ulcers will be examined on a weekly basis by a researcher with no awareness regarding the allocation of the individuals to the different groups and will assess, signs of infection, edema, redness, heat and the presence of gangrene. Photographs of the ulcers will also be taken for the subsequent determination of the area. Another researcher with no knowledge regarding the allocation of the participants will measure the surface of the ulcers with the aid of the ImageJ software program. The data will be submitted to appropriate statistical analyses. After closure of the ulcers, the patients will be followed up for a period of six months.

DETAILED DESCRIPTION:
Justification Various studies have demonstrated that phototherapy (laser or LED) is effective at enhancing skin wounds. The biological effects of both forms are similar and related to an increase in fibroblasts, the stimulation of angiogenesis, an increase in collagen synthesis, the formulation of granulation tissue and a reduction in inflammatory cells. Moreover, both forms of phototherapy increase the healed area in a shorter period of time, with LED demonstrating a late-onset effect on the healing process. In patients with partial foot amputation, this time is crucial for the fitting of the prosthetic and, consequently, the beginning of physical therapy and early locomotion. Diminishing the treatment time, with the patient observing a gradual progression in the healing process and experiencing a consequent increase in quality of life, could be a transforming factor to avoid the recurrence of ulcers and avoid further amputations.

Hypothesis

Alternative hypothesis: LED therapy is effective at potentiating the complete closure of ulcers in a shorter time following minor amputations in individuals with Diabetes mellitus.

Hull hypothesis: LED therapy is not effective at potentiating the complete closure of ulcers in a shorter time following minor amputations in individuals with Diabetes mellitus.

Methods A single-center, randomized, controlled, double-blind clinical trial with two parallel groups will be conducted in accordance with the criteria contained in the Consolidated Standards of Reporting Trials (CONSORT statement).

The sample will be composed of patients diagnosed with Diabetes mellitus in medical follow up at the vascular outpatient clinic of the Mandaqui Hospital Complex of São Paulo. Twenty patients will be analyzed in each group, as this is the estimate of surgical treatment for each vascular surgeon in a one-year period at the Mandaqui Hospital Complex.

Randomization and formation of groups Patient allocation will be performed by a researcher with no contact with the patients or main researchers. Randomization will be conducted in blocks of four for the balanced distribution of the experimental groups. For such, a lottery of 40 numbers will be conducted using a free program available at http://www.randomization.com, version from March 29, 2013.

Opaque envelopes will be identified with sequential numbers. A piece of paper containing information on the corresponding group determined through the randomization process (control or LED) will be placed into each envelope. The envelopes will remain sealed in numeric order in a secure location until the time of the treatments of the post-amputation ulcers. The researcher in charge of the randomization process and preparation of the envelopes will not be involved in any other aspect of the study.

Immediately following surgery, the main researcher, who will be in the surgical ward, will open an envelope without altering the numeric sequence and will perform the procedure indicated (active LED + bandaging or placebo LED + bandaging). The 40 patients will be allocated to the experimental and control groups in an equal fashion.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older;
* type 2 diabetes;
* either gender;
* adequate cognitive capacity to maintain the foot without load or pressure as much as possible based on the location of the ulcer;
* under care at the vascular surgery outpatient clinic of the Mandaqui Hospital Complex between January 2017 and december 2018, having undergone partial minor amputation at the same hospital (toes, foot, disarticulation at the metatarsal-phalangeal or transmetatarsal joint).

Exclusion Criteria:

* presence of infected ulcers;
* under surveillance for cancer or having undergone anti-neoplasm treatment in previous three months;
* currently pregnant or nursing;
* uncontrolled diabetes;
* Neuropathic arthropathy;
* participation in other concomitant clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Wound closure | 6 months
  The primary outcome will be the complete closure of the ulcer, which is defined as 100% epithelialization of the operated surface with no exudate, draining or need for bandages.

SECONDARY OUTCOMES:
Time for closure | up to 6 months
  time (in days) needed for complete ulcer closure.
Ulcer closure rate | up to 6 months
  On a weekly basis, the surgical wounds will be photographed with a digital camera (Canon Powershot S5 IS semi-professional, manual mode) on the upper and lower portions of the foot always at the same distance and with a millimeter scale on the left side for reading by the software program. The area of the ulcers will subsequently be measured with the aid of the ImageJ program (free software, NIH, Maryland, USA) and a software program developed by the research group for this purpose (Deana et al., 2013).
Cost-benefit ratio of ulcer treatment following minor amputations | up to 6 months
  The cost-benefit analysis will involve the determination of expenditures on materials, equipment, labor and transportation costs calculated as a function of treatment time.

CONTACTS AND LOCATIONS:
Overall Officials: Cristiane M Franca, PhD, Principal Investigator — University of Nove de Julho
Locations (1):
- Universidade Nove de Julho, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tchanque-Fossuo CN, Ho D, Dahle SE, Koo E, Li CS, Isseroff RR, Jagdeo J. A systematic review of low-level light therapy for treatment of diabetic foot ulcer. Wound Repair Regen. 2016 Mar;24(2):418-26. doi: 10.1111/wrr.12399. Epub 2016 Mar 2. PMID 26748691
- [Background] Game FL, Apelqvist J, Attinger C, Hartemann A, Hinchliffe RJ, Londahl M, Price PE, Jeffcoate WJ; International Working Group on the Diabetic Foot. Effectiveness of interventions to enhance healing of chronic ulcers of the foot in diabetes: a systematic review. Diabetes Metab Res Rev. 2016 Jan;32 Suppl 1:154-68. doi: 10.1002/dmrr.2707. PMID 26344936
- [Result] Tchanque-Fossuo CN, Ho D, Dahle SE, Koo E, Isseroff RR, Jagdeo J. Low-level Light Therapy for Treatment of Diabetic Foot Ulcer: A Review of Clinical Experiences. J Drugs Dermatol. 2016 Jul 1;15(7):843-8. PMID 27391634
- [Result] Nteleki B, Abrahamse H, Houreld NN. Conventional podiatric intervention and phototherapy in the treatment of diabetic ulcers. Semin Vasc Surg. 2015 Sep-Dec;28(3-4):172-83. doi: 10.1053/j.semvascsurg.2016.02.001. Epub 2016 Feb 18. PMID 27113284
- [Result] Cg SK, Maiya AG, Hande HM, Vidyasagar S, Rao K, Rajagopal KV. Efficacy of low level laser therapy on painful diabetic peripheral neuropathy. Laser Ther. 2015 Oct 2;24(3):195-200. doi: 10.5978/islsm.15-OR-12. PMID 26557734
- [Result] Tardivo JP, Baptista MS, Correa JA, Adami F, Pinhal MA. Development of the Tardivo Algorithm to Predict Amputation Risk of Diabetic Foot. PLoS One. 2015 Aug 17;10(8):e0135707. doi: 10.1371/journal.pone.0135707. eCollection 2015. PMID 26281044